CLINICAL TRIAL: NCT05266560
Title: Effects of Ciprofol Anesthesia on Learning and Memory Function and Antidepressant Efficacy of ECT in Patients With Depression
Brief Title: Effects of Ciprofol Anesthesia on Learning and Memory Function and Antidepressant Effects of ECT in Depressive Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, Professor.Min, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C-ECT20220214
Record Dates: First submitted 2022-02-14; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol injection group (1.5mg/kg) (Active Comparator): The patients in the propofol group were given intravenous injection of propofol 1.5 mg/kg and succinylcholine 1 mg/kg in turn, and the interval between each drug administration was 1 minute, and electroconvulsive therapy was performed after the patients were anesthetized.
  Interventions: Drug: Propofol
- Ciprofol injection group(0.4mg/kg) (Experimental): The patients in the ciprofol group were given intravenous injection of ciprofol 0.4 mg/kg and succinylcholine 1 mg/kg in turn. The interval between each drug administration was 1 minute, and the patients received electroconvulsive therapy after anesthesia.
  Interventions: Drug: ciprofol

INTERVENTIONS:
Drug: ciprofol — A new type of anesthetic drug, Ciprofol, which is newly listed and has national independent intellectual property rights, is an analogue of propofol. Its chemical name is 2-[(1R)-1-cyclopropylethyl]-6-isopropyl-phenol, and it acts on GABAA receptors like propofol. Compared with propofol, ciprofol is 4-5 times more potent, which can significantly reduce the amount of anesthetics.
  Other Names: 2-[(1R)-1-cyclopropylethyl]-6-isopropyl-phenol
  Arms: Ciprofol injection group(0.4mg/kg)
Drug: Propofol — Propofol is a commonly used anesthetic in clinical practice and is often used before ECT.
  Other Names: 2,6-Diisopropylphenol
  Arms: Propofol injection group (1.5mg/kg)

SUMMARY:
In this clinical study, propofol was used as the positive control, and a randomized controlled trial design was used to observe the effects of ciprofol anesthesia on learning and memory function and antidepressant efficacy in patients with ECT. A total of 390 depressed patients who were to undergo electroconvulsive therapy were selected and randomly divided into two groups, namely the propofol group (n=195 cases) and the ciprofol group (n=195 cases). The patients in the propofol group were given propofol 1.5mg/kg + succinylcholine 1mg/kg, and the patients in the ciprofol group were given ciprofol 0.4mg/kg and succinylcholine 1mg/kg, and the patients were given electroshock after anesthesia treat.

DETAILED DESCRIPTION:
Ciprofol injection, whose active component (HSK3486) is propofol analogue, is a novel treatment for anesthesia induction and maintenance. It has been authorized for commercialization in China on December 14, 2020.

The purpose of this experiment is to know the effect of ciprofol on the antidepressant effect and cognitive function of depressive patients after electroconvulsive therapy. Ciprofol is very similar in structure to propofol, so propofol was used as the control group in this experiment.

ELIGIBILITY:
Inclusion Criteria:

1. Depressed patients who plan to receive MECT.
2. Meet the diagnostic criteria of DSM-IV depression
3. 16≤age≤45 years old, gender is not limited
4. ASA score is I or II
5. The depressive episode lasted for at least 2 weeks
6. Clearly understand and voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Combined with serious physical diseases, such as uncontrolled hypertension, coronary heart disease, intracranial vascular malformations, asthma attacks, severe liver and kidney dysfunction, etc.
2. Foreign bodies in the body: such as pacemakers, intracranial electrodes, etc.
3. Those who have a history of epilepsy
4. Those who are taking reserpine
5. Those with acute and systemic infectious diseases, with moderate or higher fever
6. Those with a history of manic episodes
7. Those with anesthetics, Allergic to muscle relaxants
8. Pregnant women
9. Glaucoma
10. Bipolar disorder, or combined with other mental illnesses, mental retardation
11. Those who are judged not suitable for MECT treatment by the competent physician
12. History of drug abuse

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 390 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment rate within 24 hours after the whole ECT course | After the patient received MECT treatment within 24 hours after the whole ECT course
  Percentage of patients with cognitive impairment within 24 hours after the whole ECT course